CLINICAL TRIAL: NCT04828759
Title: Combining Immersive Virtual Reality With Telerehabilitation to Provide Language Intervention for People With Aphasia: A Randomized Waitlist Controlled Trial
Brief Title: Virtual Reality in Aphasia Telerehabilitation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Oulu (Other)
Collaborators: Peili Vision Oy (Unknown); Verve Oulu (Unknown); City of Oulu (Unknown)
Responsible Party: Principal Investigator, Matti Lehtihalmes, Professor, University of Oulu
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 70/2020
Record Dates: First submitted 2021-03-23; First posted 2021-04-02 (Actual); Last update posted 2021-04-02 (Actual); Status verified 2021-03

CONDITIONS: Aphasia, Acquired
Keywords: aphasia, virtual reality, head-mounted device, rehabilitation, telerehabilitation
MeSH Terms: conditions — Aphasia | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VR-treatment, then Treatment as usual (Experimental): Participants will receive 8 weeks of VR-treatment. Participants are allowed to practice as much as they wish during the VR-intervention. However, they are given a recommendation of the amount of practice (5 h / week). Before the VR-intervention, the participants will receive a guidance for using the VR-devices (i.e. orientation period) by the SLT. Participants will be able to contact the SLT freely during the 8 weeks VR-intervention period. After the orientation period, the participants will be practicing at their homes independently. However, they will receive remote guidance by the SLT. The guidance includes weekly remote guidance sessions by SLT (8 x 45 min) to ensure that training is fluent and unproblematic. Additionally, the content of exercises can be modified during these sessions. The SLT is also able to monitor the training of participants with the system. Devices: VR headset and controller, Tablet computer.
  Interventions: Behavioral: VR-treatment
- Treatment as usual, then VR-treatment (Experimental): Wait list control group: During the waitlist period the participants will receive the traditional speech and language therapy rehabilitation offered by (if offered) the general health care system in their own home municipality. The amount of rehabilitation is not controlled during the wait list period. However, the amount of received traditional speech and language rehabilitation in waitlist period will be documented. The waitlist control group will receive the same VR intervention period after the 8 weeks waitlist period.
  Interventions: Behavioral: Treatment as usual

INTERVENTIONS:
Behavioral: VR-treatment — The participants will be randomized either to group which receives the VR-intervention immediately (A) or to the waitlist control group (B). After the baseline assessment, the participants in the group A participate VR-intervention lasting for 8 weeks, and the participants in the group B will receive 8 weeks waitlist period. After the 8 weeks, the groups switch their places
  Arms: VR-treatment, then Treatment as usual
Behavioral: Treatment as usual — The participants will be randomized either to group which receives the VR-intervention immediately (A) or to the waitlist control group (B). After the baseline assessment, the participants in the group A participate VR-intervention lasting for 8 weeks, and the participants in the group B will receive 8 weeks waitlist period. After the 8 weeks, the groups switch their places
  Arms: Treatment as usual, then VR-treatment

SUMMARY:
The main purpose of this study is to evaluate the use of the immersive 3D HMD VR technology in the language intervention with a home-based telerehabilitation approach for people with aphasia. The assessments will be conducted at the baseline (prior the intervention periods) and after each intervention period (i.e. after the VR-intervention period and the waitlist period).

DETAILED DESCRIPTION:
The purpose of the present project is to study the effects, feasibility, and the participants' experiences of this novel kind of language intervention. The effects of the intervention will be studied with various outcome measures in terms of language performance, functional communication, and quality of life. The aim is to explore the VR-intervention on the group level and with a randomized waitlist control group design (or delayed crossover design). In this study, the people with aphasia will be practicing at their home with support of their relatives, and participants will also receive regular remote guidance by a speech and language therapist (SLT) during the intervention. The relatives are also involved in the assessment process.

ELIGIBILITY:
Inclusion Criteria:

* Post-stroke aphasia ≥ 3 months from stroke
* Age 18-75 years
* Finnish as a native language
* Relative have the motivation and willingness to support person with aphasia in rehabilitation process
* At least some level of spoken output
* Moderate-to-severe aphasia
* Deficit in a word retrieval process

Exclusion Criteria:

* Participation in other intervention study during the study
* Participation in other traditional speech and language therapy during the VR-intervention (i.e. 9-10 weeks period).
* Severe and current psychotic disorder
* Dementia/other neurodegenerative disease
* History of previous stroke (/strokes) if not recovered, excluding TIAs (the criteria for the recovery: no residual aphasia or other disabilities caused by stroke which would affect in significant manner on everyday life)
* Active epilepsy / migraine (< 3 years)
* Severe apraxia of speech
* Inability to act according to given instruction
* Severe neuropsychological disorder or the decline of cognitive / memory functions, which would significantly affect for training during the VR-intervention
* Vision or hearing impairment which would prevent the use of VR HMD
* if the participant's treatment or medication is unsuitable with the use of VR HMD device as assessed by the physician
* if the participant has the pacemaker or implantable (electric) medical device

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-04-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in language abilities from baseline to week 9 and to week 18 | Change from baseline to week 9 and to week 18
  Language abilities are assessed using language quotient LQ score of Western Aphasia Battery (WAB), performed at the baseline (prior the intervention periods) and after each intervention period (i.e. after the VR-intervention period and the waitlist period)
Change in naming abilities from baseline to week 9 and to week 18 | Change from baseline to week 9 and to week 18
  Naming abilities for nouns and verbs are assessed with Boston Naming Test (BNT) and TNT-test (action naming test in Finnish) performed at the baseline (prior the intervention periods) and after each intervention period (i.e. after the VR-intervention period and the waitlist period)
Change in verbal fluency from baseline to week 9 and to week 18 | Change from baseline to week 9 and to week 18
  Verbal fluency is assessed using multiple categories (produced words per one minute in each category), performed at the baseline (prior the intervention periods) and after each intervention period (i.e. after the VR-intervention period and the waitlist period)
Change in functional communication skills from baseline to week 9 and to week 18 | Change from baseline to week 9 and to week 18
  Functional communication skills are assessed with Communication Effectiveness Index (CETI), performed at the baseline (prior the intervention periods) and after each intervention period (i.e. after the VR-intervention period and the waitlist period)
Change in quality of life from baseline to week 9 and to week 18 | Change from baseline to week 8 and to week 18
  Quality of life is assessed with Stroke and Aphasia Quality of Life Scale-39 (SAQOL-39), performed at the baseline (prior the intervention periods) and after each intervention period (i.e. after the VR-intervention period and the waitlist period)

SECONDARY OUTCOMES:
Attrition rates during the study. | Through study completion, up to 18 weeks
  Amount of drop outs of participants during the study,
Participants' experiences of the VR-intervention | After VR-intervention period, at the week 9 or at the week 18, depending of the group the patient has been randomized
  The structural survey of participants' experiences of the VR-intervention.
Data collected by VR-devices regarding the performance of participants during the VR-intervention | Through the VR-intervention up to 8 weeks or through the weeks 10-17, depending of the group the patient has been randomized
  Amounts of training (in minutes) and e.g. naming speed and range of head movements collected automatically by VR-devices
Date collected by remote sessions regarding the experiences of participants and feasibility of VR-intervention | Weekly during the VR-intervention up to 8 weeks or through the weeks 10-17, depending of the group the patient has been randomized
  Data collected with semi-structural interview during remote guidance sessions (8 times during the VR-period) by the researcher. In addition, participants will be able to contact the researcher freely during the 8 weeks VR-intervention period.
Participants' experiences of the waitlist period | After waitlist period, at the week 9 or at the week 18, depending of the group the patient has been randomized
  The structural survey of participants' experiences of the waitlist period

IPD SHARING:
Plan to Share IPD: No